CLINICAL TRIAL: NCT05647902
Title: Serum Asprosin Concentrations in Patients With Periodontitis and Acute Coronary Syndrome
Brief Title: Association of Asprosin in Periodontitis and Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sema Nur Sevinc, Assistant Professor, Ataturk University
Other Study IDs: MIC3
Record Dates: First submitted 2022-12-04; First posted 2022-12-13 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Diseases; Periodontal Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Group: 70 systemically healthy patients; 35 healthy gingiva is divided into 2 subgroups, 35 of which are periodontitis. Asprosin levels will be examined biochemically in serum samples taken from patients.
  Interventions: Diagnostic Test: Serum samples will be collected. Asprosin levels will be determined by biochemical analysis
- Myocard Infactus Group: 50 patients with myocardial infarction; 25 healthy gingiva is divided into 2 subgroups, 25 of which are periodontitis. Asprosin levels will be examined biochemically in serum samples taken from patients.
  Interventions: Diagnostic Test: Serum samples will be collected. Asprosin levels will be determined by biochemical analysis

INTERVENTIONS:
Diagnostic Test: Serum samples will be collected. Asprosin levels will be determined by biochemical analysis — Serum samples will be collected from both groups for biochemical analysis.

SUMMARY:
Asprosin, a recently discovered glucogenic adipokine, is mainly synthesized by white adipose tissue and released during fasting. Appetite, glucose metabolism, insulin resistance, cell apoptosis, etc. asprosin is associated with diseases such as diabetes, obesity, polycystic ovary syndrome, and cardiovascular diseases. Periodontal tissue may act as a source of endocrine-like inflammatory mediators (such as TNF-α, IL-6 and IL-1) that are important in periodontal inflammation and can affect glucose and lipid metabolism. Production of TNF-α and IL-6 in adipose tissues strengthens the relationship between cardiovascular diseases and periodontitis. Investigators postulated that asprosin may be a candidate for explaining the triangular relationship between cardiovascular and periodontal disease.

DETAILED DESCRIPTION:
Periodontal disease is a chronic, multifactorial, and infectious disease caused by bacteria. It is characterized by the formation of an inflammatory response in the supporting bone and connective tissue against microbial dental plaque, and the nature of the resulting inflammatory response determines the course of periodontal disease. Cardiovascular and periodontal diseases are closely related, presenting a triad association. Asprosin circulates in the blood at nanomolar levels and is taken to the liver, where it activatesinvestigators the G protein-cAMP-PKA pathway, causing rapid glucose release into the circulation.

ELIGIBILITY:
Inclusion Criteria:

For Healthy group

* All individuals were generally healthy,
* non-smoking For Myocard Infarctus group
* patients with ST elevation of Myocardial Infactus
* patient with less than ten teeth

Exclusion Criteria:

* Smokers or those with diabetes or other inflammatory disease
* Pregnant or breastfeeding women
* None had undergone periodontal therapy and/or antibiotic therapy in the past 6 months.
* None has a contagious disease such as HIV or AIDS

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was carried out on 120 patients, 50 admitted to Atatürk University Medical Faculty Heart Center with SD elevation myocardial infarction and 70 who applied to Atatürk University Faculty of Dentistry. Patients who consent to participate in the study on a randomized basis and comply with the inclusion criteria are divided into periodontitis and healthy groups after the periodontal examination. Body mass index was evaluated
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Asprosin Levels | two weeks
  Determination of asprosin levels by making biochemical analyzes from serum

CONTACTS AND LOCATIONS:
Overall Officials: Oğuzhan Birdal, Asist. Prof., Study Chair — Ataturk University
Locations (1):
- Atatürk University Faculty of Dentistry, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Romere C, Duerrschmid C, Bournat J, Constable P, Jain M, Xia F, Saha PK, Del Solar M, Zhu B, York B, Sarkar P, Rendon DA, Gaber MW, LeMaire SA, Coselli JS, Milewicz DM, Sutton VR, Butte NF, Moore DD, Chopra AR. Asprosin, a Fasting-Induced Glucogenic Protein Hormone. Cell. 2016 Apr 21;165(3):566-79. doi: 10.1016/j.cell.2016.02.063. Epub 2016 Apr 14. PMID 27087445
- [Result] Yuan M, Li W, Zhu Y, Yu B, Wu J. Asprosin: A Novel Player in Metabolic Diseases. Front Endocrinol (Lausanne). 2020 Feb 19;11:64. doi: 10.3389/fendo.2020.00064. eCollection 2020. PMID 32153505